CLINICAL TRIAL: NCT05583357
Title: A Single Center, Randomized, Open-labeled, Blind Endpoint Evaluation, Exploratory Clinical Study to Evaluate the Safety and Immunogenicity of Bivalent Vaccine V-01D-351 as a Booster Dose in Participants Aged 18 Years and Older Vaccinated 2-dose or 3-dose Inactivated COVID-19 Vaccine
Brief Title: Exploratory Clinical Study to Evaluation of the Safety and Immunogenicity of Bivalent Vaccine V-01D-351
Acronym: COVID-19
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: V-01D-351-Booster-03
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental)
  Interventions: Biological: V-01D-351
- Cohort 2 (Experimental)
  Interventions: Biological: V-01D-351
- Cohort 3 (Active Comparator)
  Interventions: Biological: CoronaVac
- Cohort 4 (Active Comparator)
  Interventions: Biological: CoronaVac

INTERVENTIONS:
Biological: V-01D-351 — One dose of V-01D-351 on participants received 2 doses of inactivated vaccine (CoronaVac) 6-15 months ago
  Arms: Cohort 1
Biological: V-01D-351 — One dose of V-01D-351 on participants received 3 doses of inactivated vaccine (CoronaVac) 5-9 months ago
  Arms: Cohort 2
Biological: CoronaVac — One dose of CoronaVac on participants received 2 doses of inactivated vaccine (CoronaVac) 6-15 months ago
  Arms: Cohort 3
Biological: CoronaVac — One dose of CoronaVac on participants received 3 doses of inactivated vaccine (CoronaVac) 5-9 months ago
  Arms: Cohort 4

SUMMARY:
It is a single center, randomized, open-labeled, blind endpoint evaluation, exploratory clinical study to evaluate the safety and immunogenicity of bivalent vaccine V-01D-351 as a booster.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older at time of consent, male or female;
* Normal body temperature;
* Meet either of the following conditions:

  1. Received completed primary immunization of 2 doses of CoronaVac 6-15 months ago;
  2. Received completed 3 doses of CoronaVac 5-9 months ago;
* Female participants who are not pregnant at the time of enrollment (urine pregnancy test is negative), nor during lactating; and has no birth plan and agree to take effective contraception in 7 months after enrollment; and took effective and acceptable contraceptive methods in the previous 2 weeks before the enrollment;
* Be able and willing to complete the study during the entire study and follow-up period;
* Participants who have the ability to understand the study process, sign the informed consent form voluntarily , and be able to comply with the requirements of the clinical study protocol.

Exclusion Criteria:

* Serious chronic diseases or uncontrolled diseases;
* Uncontrolled neurological disorders, epilepsy;
* Received any inactivated vaccine within 1 week or received any attenuated vaccines within 4 weeks;
* Patients with congenital or acquired immunodeficiency;
* History of severe allergy or be allergic to any components of the test vaccines;
* History of hereditary hemorrhagic tendency or coagulation dysfunction;
* Patients with malignant tumors and other patients have a life expectancy less than 1 year;
* Refuse to sign the informed consent form or inability to complete follow-ups as required by the protocol;
* History of previous COVID-19 infection;
* Pregnant or breastfeeding women, or females of childbearing potential who not agree to or able to take effective and acceptable contraceptive methods during the study;
* Participants who have participated in other clinical trials within 3 months or are participating in other clinical trials;
* Those considered by the investigator as inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
Neutralizing antibody GMT of Omicron BA.5 | 28 days after vaccination
  Neutralizing antibody GMT of the most prevalent SARS-CoV-2 variant (Omicron BA.5)

SECONDARY OUTCOMES:
Neutralizing antibody GMT of other SARS-CoV-2 variants | 7 days, 14 days, 28 days, 3 months, 6 months and 12 months after vaccination
  Neutralizing antibody GMT of Delta variant and Omicron variants (BA.2, BA.4, BA.5)
Neutralizing antibody titer of other SARS-CoV-2 variants (MRNT) | 7 days, 14 days, 28 days, 3 months, 6 months and 12 months after vaccination
  Neutralizing antibody titer of Delta variant and Omicron variants (BA.2, BA.4, BA.5) by MRNT
Neutralizing antibody titer of other SARS-CoV-2 variants (SVNT) | 7 days, 14 days, 28 days, 3 months, 6 months and 12 months after vaccination
  Neutralizing antibody titer of Delta variant and Omicron variants (BA.2, BA.4, BA.5) by SVNT
Total IgG antibody level | 7 days, 14 days, 28 days, 3 months, 6 months and 12 months after vaccination
  Total IgG antibody level of SARS-CoV-2
Spike protein antibody level | 7 days, 14 days, 28 days, 3 months, 6 months and 12 months after vaccination
  Antibody level of anti-SARS-CoV-2 spike protein
RBD antibody level | 7 days, 14 days, 28 days, 3 months, 6 months and 12 months after vaccination
  Anti-SARS-CoV-2 RBD antibody level
Specific cytokine secretion levels | 7 days, 14 days, 28 days, 3 months, 6 months and 12 months after vaccination
  Specific cytokine secretion levels such as IFN-γ
AEs | 30 minutes, 0-7 days, 0-28 days after vaccination
  Observe the AEs occurs at different time point after vaccination
SAE and AESI | Within 12 months after vaccination
  Observe the SAE and AESI after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoguan Hospital of Chinese Medicine, Shaoguan, Guangdong, China